CLINICAL TRIAL: NCT01152671
Title: A Multiple Center Randomized, Double-Blind, Single-Ascending-Dose, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics Following Oral Administration of RO5024048 in Healthy Japanese and Caucasian Subjects
Brief Title: A Study of RO5024048 in Japanese and Caucasian Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PP25311
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: RO5024048
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — single oral dose
  Arms: Arm 2
Drug: RO5024048 — single oral dose
  Arms: Arm 1

SUMMARY:
This randomized, double-blind, placebo-controlled study will assess the safety, tolerability and pharmacokinetics of RO5024048. Japanese and Caucasian healthy volunteers will be randomized to receive either single oral doses of RO5024048 or placebo. Follow-up is 7-10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, 20 to 55 years of age, inclusive
* Body mass index (BMI) 18 - 30 kg/m2 inclusive
* Non-smoker, or previous smoker who discontinued smoking >/= 6 month prior to study entry
* Japanese subjects must be first generation: born in Japan, not having lived outside Japan >5 years, able to trace maternal and paternal Japanese ancestry
* Female subjects of childbearing potential and male subjects and their partners of childbearing potential must agree to use two forms of contraception
* Agree to abstain from alcohol consumption and from strenuous exercise up to 3 days before dosing and throughout study (including the follow-up visit)

Exclusion Criteria:

* Positive pregnancy test
* Males whose female partner is pregnant or trying to become pregnant
* Positive urine test for drugs of abuse
* Positive for alcohol
* Positive result on hepatitis B, hepatitis C, or HIV test
* Clinically significant disease or abnormalities in laboratory parameters
* Participation in an investigational drug, biologic or device study within 3 months before study drug administration
* Donation or loss of any blood over 450 mL within 3 months before study drug administration

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2010-06; Study Completion 2010-08

PRIMARY OUTCOMES:
Pharmacokinetics of RO4995855 (parent of the prodrug RO5024048) and its metabolite(s) | Day 1 to Day 4

SECONDARY OUTCOMES:
Safety and tolerability: Adverse events, laboratory parameters, ECG | Day 1 to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Glendale, California
  - Eatontown, New Jersey